CLINICAL TRIAL: NCT04087291
Title: VERDICT (Veterans Response to Dosage in Chiropractic Therapy): A Pragmatic Randomized Trial Addressing Dose Effects for Chronic Low Back Pain
Brief Title: Veterans Response to Dosage in Chiropractic Therapy
Acronym: VERDICT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palmer College of Chiropractic (Other)
Collaborators: Yale University (Other); University of Iowa (Other); Dartmouth College (Other); VA Connecticut Healthcare System (U.S. Federal Agency); Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency); Iowa City VA Health Care System (U.S. Federal Agency); VA Greater Los Angeles Healthcare System (U.S. Federal Agency); Office of Research on Women's Health (ORWH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 18-34; UH3AT009761 (NIH)
Record Dates: First submitted 2019-08-27; First posted 2019-09-12 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Low Back Pain; Patient Acceptance of Health Care; Veterans Health
Keywords: chronic; pain management; manipulation, chiropractic
MeSH Terms: conditions — Low Back Pain; Patient Acceptance of Health Care; Bronchiolitis Obliterans Syndrome; Agnosia | interventions — Manipulation, Chiropractic

STUDY DESIGN:
Intervention Model Description: This pragmatic, parallel groups, multisite randomized trial will include Veterans with cLBP who will be randomly allocated to undergo a course of a low dose (1-5 visits) or a higher dose (8-12 visits) of multimodal, evidence-based chiropractic care for 10 weeks (Phase 1). Group allocation will occur through a 1:1 ratio by a predetermined, computer-generated, restricted randomization scheme with random block sizes, stratified by site and sex. After Phase 1, participants within each treatment arm will be randomly allocated again to receive either chiropractic chronic pain management (CCPM) consisting of scheduled monthly chiropractic care or no CCPM for 10 months. This second group allocation will also occur through a 1:1 ratio to Phase 2 within low dose or higher dose in Phase 1 by a predetermined, computer-generated, restricted randomization scheme with random block sizes, stratified by site and sex.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Doctors of Chiropractic (DCs), site study coordinators (SCs), participants and interviewers will not be blinded to treatment group assignment; DCs will not see research outcome measures; statisticians will be blinded to treatment group assignment during data analysis; and research personnel conducting Computerized Adaptive Testing Interviews (CATIs) will be blinded to study group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase 1: Low Dose (1-5 visits) (Active Comparator): Veterans with cLBP who will be randomly allocated to undergo a course of a low dose (1-5 visits) of multimodal, evidence-based chiropractic care for 10 weeks (Phase 1).
  Interventions: Other: Chiropractic Care
- Phase 1: Higher Dose (8-12 visits) (Active Comparator): Veterans with cLBP who will be randomly allocated to undergo a course of a higher dose (8-12 visits) of multimodal, evidence-based chiropractic care for 10 weeks (Phase 1).
  Interventions: Other: Chiropractic Care
- Phase 2: CCPM (Active Comparator): After Phase 1, Veterans with cLBP who will be randomly allocated again to receive chiropractic chronic pain management (CCPM) consisting of scheduled monthly chiropractic care for 10 months.
  Interventions: Other: Chiropractic Care
- Phase 2: No CCPM (No Intervention): After Phase 1, Veterans with cLBP who will be randomly allocated again to receive no CCPM in which they will receive no chiropractic care for 10 months.

INTERVENTIONS:
Other: Chiropractic Care — Chiropractic interventions:
  1. Patient education.
  2. Passive interventions, such as spinal manipulation and myofascial therapies which include thrust type (high velocity-low amplitude) spinal manipulation for the low back, non-thrust manipulation (joint mobilization), and use of manually held instruments, such as an Activator. Myofascial therapies are also commonly used, such as myofascial release and trigger point therapy.
  3. Transitional interventions, such as therapeutic exercise.
  4. Recommendations for active interventions, such as general exercise and mind-body therapies.
  5. Self-management advice, which refers to advice given to build the capacity of a person to self-monitor, control, and/or reduce the impact of a condition over time.
  Other Names: Manipulation, Chiropractic
  Arms: Phase 1: Higher Dose (8-12 visits); Phase 1: Low Dose (1-5 visits); Phase 2: CCPM

SUMMARY:
This study evaluates how Veterans with chronic low back pain (cLBP) respond to varying doses of chiropractic therapy and how health services utilization are impacted as a result.

There are 2 phases in this study. In Phase 1, half of participants will receive a low dose (1-5 visits) of chiropractic care for 10 weeks, while the other half will receive a higher dose (8-12 visits) for 10 weeks. At the end of Phase 1, participants in each group will be randomized again to receive either chronic chiropractic pain management (CCPM) (1 scheduled chiropractic visit per month x 10 months) or no CCPM for 10 months.

DETAILED DESCRIPTION:
The combination of chronic low back pain (cLBP) and high medication use negatively impacts Veterans' work productivity and quality of life, and generates substantial risk for long-term disability and opioid addiction. Although non-pharmacological therapies, such as those commonly used by doctors of chiropractic (DCs), are recommended by recent guidelines for treatment of cLBP, the optimal patterns of chiropractic use, clinical impact of chiropractic treatment on other health services utilization, and long-term effectiveness of chiropractic care is unknown.

This is a pragmatic, parallel groups, multisite randomized trial. Veterans with cLBP are randomly allocated to undergo a course of a low dose (1-5 visits) or a higher dose (8-12 visits) of multimodal, evidence-based chiropractic care for 10 weeks (Phase 1). The investigators hypothesize that a higher dose (8-12 visits) of chiropractic care will be more effective in improving function and reducing pain intensity and pain-related interference in Veterans with cLBP compared to a low dose (1-5 visits).

After Phase 1, participants within each treatment arm will be randomly allocated again to receive either chronic chiropractic pain management (CCPM) consisting of scheduled monthly chiropractic care or no CCPM for 10 months. The investigators hypothesize that CCPM (1 scheduled chiropractic visit per month x 10 months) will result in improved function, and reduced pain intensity, pain-related interference, and average number of days per week with low back pain (LBP) in Veterans with cLBP compared to no CCPM.

This study will also evaluate the impact of CCPM on health services outcomes compared to no CCPM. Evaluation of health services utilization at 52 weeks will include use of prescription medications, including opioids, referrals and number of visits to other healthcare professionals or service lines (physical therapy, injections, surgery, etc.), and hospitalizations for any cause and for cLBP.

Finally, the investigators will evaluate patient and clinician perceptions of non-specific treatment factors, effectiveness of study interventions, and impact of the varying doses of standard chiropractic care and the CCPM on clinical outcomes across 4 VA facilities using a mixed method, process evaluation approach.

ELIGIBILITY:
Inclusion Criteria:

* Veterans aged ≥ 18 years
* Self-reported cLBP
* Has low back related pain and disability
* Able to comprehend study details without need for a proxy
* Diagnostic confirmation of neuromusculoskeletal LBP
* Willing and able to attend up to 1 year of outpatient chiropractic visits

Exclusion Criteria:

* Any condition prohibiting or contraindicating chiropractic care
* Inability to complete outcomes and/or provide informed consent as determined by the site SC during the consent process
* Established plans to move within 3 months
* Under active chiropractic care
* No phone
* No email address
* Participating in another study investigating treatment(s) for pain
* Current or planned hospice care
* Current or planned pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 766 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Low Back Pain Disability at several time points - Roland Morris Disability Questionnaire (RMDQ) | At Baseline and Weeks 5, 10, 26, 40, and 52
  A one-page, 24-item questionnaire related to low back pain disability. The RMDQ can discriminate between different forms of treatment for back pain, and is sensitive to clinical change.

SECONDARY OUTCOMES:
Healthcare Services Utilization | 52 weeks
  We will assess all healthcare services used by each participant during the study period including the clinics seen, number of visits, orders, investigations, and prescriptions. We will estimate costs for these services using Decision Support System69 data. We will assess differences in cLBP-related healthcare utilization in the 4 treatment groups (low dose-CCPM, low dose-no CCPM, higher dose-CCPM, higher dose-no CCPM). In addition, we will investigate differences in health care utilization between sites.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Goertz, DC, PhD, Principal Investigator — Duke University; Cynthia Long, PhD, Principal Investigator — Palmer Center for Chiropractic Research (PCCR)
Locations (4):
- United States (4):
  - VA Greater Los Angeles Health Care System, Los Angeles, California
  - VA Connecticut Healthcare System, West Haven, Connecticut
  - Iowa City VA Health Care System, Iowa City, Iowa
  - Minneapolis VA Health Care System, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No
Depending upon the needs and desires of the requesting party, the data that are shared may include analytic tables or de-identified, limited data sets that are transmitted to the requesting parties for additional analyses. In order to safeguard patient confidentiality and scientific integrity, the investigators will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) evidence of local IRB approval from the requesting party's home institution; (2) a commitment to use the data only for research purposes and not to identify any individual participant; (3) a commitment to secure the data using appropriate computer technology to protect the privacy and security of the individual participant; (4) a commitment to destroy or return the data after analyses are completed; and (5) an assurance to use the data in compliance with all applicable statutes and regulations, including but not limited to the HIPAA.

REFERENCES:
- [Background] Long CR, Lisi AJ, Vining RD, Wallace RB, Salsbury SA, Shannon ZK, Halloran S, Minkalis AL, Corber L, Shekelle PG, Krebs EE, Abrams TE, Lurie JD, Goertz CM. Veteran Response to Dosage in Chiropractic Therapy (VERDICT): Study Protocol of a Pragmatic Randomized Trial for Chronic Low Back Pain. Pain Med. 2020 Dec 12;21(Suppl 2):S37-S44. doi: 10.1093/pm/pnaa289. PMID 33313732
- [Background] Lisi AJ, Salsbury SA, Hawk C, Vining RD, Wallace RB, Branson R, Long CR, Burgo-Black AL, Goertz CM. Chiropractic Integrated Care Pathway for Low Back Pain in Veterans: Results of a Delphi Consensus Process. J Manipulative Physiol Ther. 2018 Feb;41(2):137-148. doi: 10.1016/j.jmpt.2017.10.001. PMID 29482827
- [Derived] Salsbury SA, Long CR, McCarey J, Lisi AJ, Steward A, Wallace RB, Goertz CM. Age differences in demographic and clinical characteristics among veterans with chronic low back pain: a cross-sectional study of baseline findings from the Veteran Response to Dosage in Chiropractic Therapy (VERDICT) trial. Chiropr Man Therap. 2025 Oct 13;33(1):44. doi: 10.1186/s12998-025-00613-z. PMID 41084026
- See also: Chiropractic Integrated Care Pathway for Low Back Pain in Veterans: Results of a Delphi Consensus Process — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6103526/
- See also: Veteran Response to Dosage in Chiropractic Therapy (VERDICT): Study Protocol of a Pragmatic Randomized Trial for Chronic Low Back Pain — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7734654/

DOCUMENTS (1):
  • Informed Consent Form (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT04087291/ICF_000.pdf